CLINICAL TRIAL: NCT04945837
Title: Psychologic Impact of COVID-19 Pandemic on the Hospital Staff of the Nouvelle Aquitaine Area : a Prospective Longitudinal Study by Self-administered Questionnaires
Brief Title: Psychologic Impact of COVID-19 Pandemic on the Hospital Staff of the Nouvelle Aquitaine Area
Acronym: IMPSY-COV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Collaborators: Regional Health Agency New Aquitaine (Other Government); Région Nouvelle Aquitaine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A02592-37
Record Dates: First submitted 2021-06-21; First posted 2021-06-30 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Personnel, Hospital; Work-Related Condition; Work-Related Stress Disorder
Keywords: COVID-19; Mental health; Anxiety; Hospital personnel; Longitudinal; Pandemic
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective Longitudinal Study by Self-administered Questionnaires
Masking Description: Data anonymisation:
  Participant timepoints data are identified and followed up through a token number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unique study arm (Other): Initial socio-demographic questionnaire 5 timepoints psychologic and self-administered questionnaires
  Interventions: Other: self administered questionnaire

INTERVENTIONS:
Other: self administered questionnaire — longitunidal descriptive study

SUMMARY:
Evaluation of the psychological impact of the COVID-19 pandemic on hospital staff in the French Nouvelle Aquitaine area, through a longitudinal study with repeated self-administered psychologic scales

DETAILED DESCRIPTION:
Evaluation of the psychological impact of Coronavirus disease 2019 (COVID-19) on hospital personnel in Nouvelle Aquitaine. IMPSY-COV Upon recent outbreaks of new diseases (SARS, MERS-CoV, Ebola) have led to the emergence of psychiatric disorders in healthcare workers , such as post-traumatic stress , anxiety (e.g., panic attacks) or depressive episodes. Observed similarities in between propagation patterns of SARS-CoV-2 and SARS, alow us to expect the occurence of similar psychiatric disorders in COVID-19 context to those described (Vignaud, Prieto, 2020). The study is set up to assess the psychological state of hospital personnel in the working conditions of treating COVID-19 suffering patients.

87000 hospital staff workers from the Nouvelle Aquitaine region will be invited to take part in the study. This includes medical and non-medical professionals from general and psychiatric hospitals exposed to COVID-19.

Study design. The protocol shows two phases and five measurement timepoints. In the initial phase (T0), eligible persons will be contacted via email. Those wishing to participate will then consent, answer socio-demographic questions and a series of psychology questionnaires. In the longitudinal phase, participants will be again invited to answer the same series of questionnaires four times: one month after the initial phase (T1), 3 months after (T2), 6 months after (T3) and 12 months after (T4).

Statistical analysis. In order to identify the consequences generated by COVID-19 in hospital personnel through a longitudinal protocol, several statistical analyses are considered, including logistic and linear regressions as well as ANOVA and MANOVA.

Expected outcomes. The study will assess the occurrence and the evolution of psychological distress and identify vulnerability factors that may trigger psychiatric disorders in these situations. The study will also provide an opportunity to improve the supporting actions of professionals affected by the crisis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* hospital workers exposed to COVID-19
* consented to participate to the study
* master the french langage
* Understanding of type, objectives and study methology
* accept an on-line evaluation
* Benefit from health insurance

Exclusion Criteria:

* refuse to participate
* pregnant or breastfeeding woman
* Be under measure of legal protection: guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in anxiety disorder overcome | inclusion, month 1, month 3, month 6, month 12
  GAD-7 score:
  > 7 , the anxiety disorder status is "supected", [5; 9] corresponds to anxiety evaluation: "light" [10; 14] corresponds to anxiety evaluation: "moderate" > 15, corresponds to anxiety evaluation: "severe"
Changes in anxiety disorder overcome | inclusion, month 1, month 3, month 6, month 12
  PDSR verifies that maximum of the panic state is reached within ten minutes

SECONDARY OUTCOMES:
Determination and collection of lived traumatic events types | inclusion, month 1, month 3, month 6, month 12
  Life Events Checklist for DSM-5 (LEC-5)
Posttraumatic stress disorder symptoms presence and measurment | inclusion, month 1, month 3, month 6, month 12
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) PCL-5 score > 32 indicate presence of Posttraumatic Stress Trouble (PST)
2-last-week mood assessment | inclusion, month 1, month 3, month 6, month 12
  Beck Depression Inventory - Fast Screen - France (BDI-FS FR) score > 13 indicates presence of a depressive trouble
Identification of coping pattern to stress | inclusion, month 1, month 3, month 6, month 12
  Coping Inventory for Stressful Situations (CISS) questionnaire Participant assess from 'little" to "a lot" his tendency to adopt a task, emotion or behaviour based pattern
Burn out diagnosis | inclusion, month 1, month 3, month 6, month 12
  MASLACH BURNOUT INVENTORY (MBI questionnaire) assessment of the 3 aspects from low to high
  * burn out feeling
  * deshumanisation
  * accomplishment at work
Self evaluation of state of health | inclusion, month 1, month 3, month 6, month 12
  considering the 4-last-weeks the participant will assess 8 under-scales for score 0 to 100 (favourable)
Psycho active drugs intakes and level of intake over the last month | inclusion, month 1, month 3, month 6, month 12
  selection of the drug and level of intake will n*be assessed 'none', "new", "increasing", constant"
Evaluation of the CUMP support to health professionnals | inclusion, month 1, month 3, month 6, month 12
  answer "yes' or "no" support has been contacted already or since the last study assessement

IPD SHARING:
Plan to Share IPD: No
Actually no sharing expected

REFERENCES:
- [Background] Chua SE, Cheung V, Cheung C, McAlonan GM, Wong JW, Cheung EP, Chan MT, Wong MM, Tang SW, Choy KM, Wong MK, Chu CM, Tsang KW. Psychological effects of the SARS outbreak in Hong Kong on high-risk health care workers. Can J Psychiatry. 2004 Jun;49(6):391-3. doi: 10.1177/070674370404900609. PMID 15283534
- [Background] Greenberg N, Docherty M, Gnanapragasam S, Wessely S. Managing mental health challenges faced by healthcare workers during covid-19 pandemic. BMJ. 2020 Mar 26;368:m1211. doi: 10.1136/bmj.m1211. No abstract available. PMID 32217624
- [Background] Johnson EI, Grondin O, Barrault M, Faytout M, Helbig S, Husky M, Granholm EL, Loh C, Nadeau L, Wittchen HU, Swendsen J. Computerized ambulatory monitoring in psychiatry: a multi-site collaborative study of acceptability, compliance, and reactivity. Int J Methods Psychiatr Res. 2009;18(1):48-57. doi: 10.1002/mpr.276. PMID 19195050
- [Background] Luceno-Moreno L, Talavera-Velasco B, Garcia-Albuerne Y, Martin-Garcia J. Symptoms of Posttraumatic Stress, Anxiety, Depression, Levels of Resilience and Burnout in Spanish Health Personnel during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Jul 30;17(15):5514. doi: 10.3390/ijerph17155514. PMID 32751624
- [Result] Mohammed A, Sheikh TL, Poggensee G, Nguku P, Olayinka A, Ohuabunwo C, Eaton J. Mental health in emergency response: lessons from Ebola. Lancet Psychiatry. 2015 Nov;2(11):955-7. doi: 10.1016/S2215-0366(15)00451-4. No abstract available. PMID 26544738
- [Result] Chan AO, Huak CY. Psychological impact of the 2003 severe acute respiratory syndrome outbreak on health care workers in a medium size regional general hospital in Singapore. Occup Med (Lond). 2004 May;54(3):190-6. doi: 10.1093/occmed/kqh027. PMID 15133143